CLINICAL TRIAL: NCT06420648
Title: A Randomized Controlled Trial Comparing Controlled Active Motion and Early Passive Mobilization Protocols for Rehabilitation of Repaired Flexor Tendons in Zone II
Brief Title: Controlled Active Motion vs Early Passive Mobilization for Flexor Tendons Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, principal investigator, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2024- 366
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Flexor Tendon Rupture

STUDY DESIGN:
Intervention Model Description: 2 arm randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early passive mobilization group (Experimental): The modified Kleinert protocol will be used as an EPM procedure. Within 3 to 5 days following surgery, the affected hand will be placed inside the dorsal slab Kleinert splint with the wrist in 30-40 flexion; metacarpophalangeal joint (MP) in 60-70-degree flexion; PIP and DIP joints in extension. Rubber band traction will be directed to the fingernail from the wrist, with a palmar pulley system. All patients will perform passive flexion and active extension exercises with an active hold for 2-3 seconds 10 times per hour. Traction will be removed at the end of 3rd week and very gentle active flexion will start at the 4th week. The splint will be removed in the 5th-6th weeks. Blocking exercises will be started at 7th-8th weeks and resisted exercises will be started after the 8th week with the full function permitted by week 12th week .
  Interventions: Other: Early passive mobilization
- Controlled active motion group (Experimental): A modified CAM protocol will be used. Exercises will be performed hourly for 10 repetitions in the form of passive flexion and active extension exercises with an active hold of the fingers in the flexed position for 2-3 seconds.
  Interventions: Other: Controlled active motion

INTERVENTIONS:
Other: Early passive mobilization — a rehabilitation protocol for post-surgical repair of flexor tendons of the hand
  Other Names: modified Kleinert protocol
  Arms: Early passive mobilization group
Other: Controlled active motion — a rehabilitation protocol for post-surgical repair of flexor tendons of the hand
  Arms: Controlled active motion group

SUMMARY:
a randomized controlled trial tends to compare 2 rehabilitation approaches - early passive mobilization (EPM) and controlled active motion (CAM) - that are commonly used in the treatment of post-surgical flexor tendon repair of the hand

DETAILED DESCRIPTION:
a randomized controlled trial tends to compare 2 rehabilitation approaches commonly used in the treatment of post-surgical flexor tendon repair of the hand. in this study, the authors try to fill the gap in the literature regarding the more effective approach. the comparisons between both approaches were scarce in previous literature.

Participants will be randomly allocated to one of two treatment groups: early passive mobilization (EPM) using a modified Kleinert protocol or controlled active motion (CAM) using a modified Duran technique (n=20). Patients were assessed at baseline and then at the 6th and 12th weeks of interventions to quantify total active motion (TAM) of the proximal and distal interphalangeal joints using goniometry, and grip strength with dynamometry. the disability level will be assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* males or females
* between 25-50 years
* Post-surgical repair of the flexor digitorum profundus (FDP) and superficialis (FDS) tendons of a single-digit
* the case should be recent (2-3 days post-surgical)

Exclusion Criteria:

* age below 25 or above 50
* a systemic disease affecting hand joints such as rheumatic arthritis
* thumb flexor tendon repair will be excluded
* chronic cases
* concurrent injuries such as phalangeal fractures, joint injuries, or significant skin loss

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Total active motion (TAM) | at baseline
  Active range of motion in proximal interphalangeal joint (PIP) and the distal interphalangeal joint (DIP) of the injured digits will be measured by manual hand goniometry. Outcome will be expressed by Strickland formula. TAM (%) = (Active flexion of PIP+DIP) - Extension Lag of both joints/175× 100 This formula can determine the percentage of recovery of TAM. The results of TAM (%) are classified in four categories: "Excellent, good, fair, and poor"
Total active motion (TAM) | after the 12th week of intervention
  This formula can determine the percentage of recovery of TAM. The results of TAM (%) are classified in four categories: "Excellent, good, fair, and poor" This formula determined the percentage of recovery of TAM. The results of TAM (%) were classified in four categories: "Excellent, good, fair, and poor"
handgrip strength | baseline
  Hand dynamometer (Jammer dynamometer) will be used to evaluate hand grip strength. Measurements will be taken for both hands for three times. The mean of three trials will be taken for every measurement occasion. The mean value in the injured hand will be expressed as percentage of the mean value in the non-injured hand as follows:
  % of hand grip strength = Mean grip strength in the involved hand/ Mean grip strength in the uninvolved hand × 100.
handgrip strength | after the 12th week of intervention
  Hand dynamometer (Jammer dynamometer) will be used to evaluate hand grip strength. Measurements will be taken for both hands for three times. The mean of three trials will be taken for every measurement occasion. The mean value in the injured hand will be expressed as percentage of the mean value in the non-injured hand as follows:
  % of hand grip strength = Mean grip strength in the involved hand/ Mean grip strength in the uninvolved hand × 100.
Functional disability | at baseline
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to measure the functional disabilities. It is a valid questionnaire used in a number of other disabling conditions of the hand. A DASH-questionnaire score, ranges from 0 to 100. A score of 0 means no difficulties in daily living and a score of 100 means maximum difficulties in performing tasks of daily living
Functional disability | after the 12th week of intervention
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire will be used to measure the functional disabilities. It is a valid questionnaire used in a number of other disabling conditions of the hand. A DASH-questionnaire score, ranges from 0 to 100. A score of 0 means no difficulties in daily living and a score of 100 means maximum difficulties in performing tasks of daily living

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Hail University Poly Clinic, Hail
  - Hisham Hussein, Hail

IPD SHARING:
Plan to Share IPD: No
data will be available with the senior author upon request